CLINICAL TRIAL: NCT04843618
Title: Prevalence and Risk Factors of Pressure Ulcers in Hospitalized Patients in Beni Suef Governorate of Egypt
Brief Title: Prevalence and Risk Factors of Pressure Ulcers in Beni Suef Governorate of Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Mahmoud Mohamed, prevalence and risk factors of pressure ulcers in hospitalized patients in Beni Suef governorate of Egypt, Cairo University
Other Study IDs: pressure ulcers
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the study aims at examining the relation between the prevalence and risk factors of pressure ulcers among hospitalized patients in Beni Suef governorate of Egypt

DETAILED DESCRIPTION:
pressure ulcers are defined as localized damage to the skin as well as underlying soft tissue, usually occuring over a bony prominence or to medical devices.

immobility and friction are important risk factors for pressure ulcers, Malnutrition and body mass index are associated with pressure injury prevalence, the days in hospital, skin moisture and other neurological factors are significant risk factors for pressure ulcer development.

Beni-Suef is one of the upper Egypt governorates located about 120 Km south of cairo, according to population estimates from 2019, the majority of residents in the governorate live in rural areas, with an urbanization rate of only 23.2%, Due to greater reliance on federal and state payers, low volume and complxity of services provided, rural residents often encounter barriers to healthcare that limit their ability to obtain the care they need

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients will be selected from ICU and CCU
* both sexes males and females
* their age ranges between 25-65 years old
* patients who have peripheral arterial disease
* their body mass index (class II and class III obesity)
* diabetic patients more than 5 years old

Exclusion Criteria:

* medically unstable patients
* un cooperative patients
* semi- conscious or unconscious patients according to glascow coma scale

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cross-sectional study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
examine the relation between the prevalence and risk factors of pressure ulcers among hospitalized patients in Beni Suef governorate of Egypt | baseline
  correlate between the prevalence and risk factors of pressure ulcers by using : sociodemographic variables, Braden risk scale assessment, clinical charactristics of the patient illness amd physical examination to assess the grade of pressure ulcer

REFERENCES:
- [Result] Bergstrom N, Horn SD, Rapp M, Stern A, Barrett R, Watkiss M, Krahn M. Preventing Pressure Ulcers: A Multisite Randomized Controlled Trial in Nursing Homes. Ont Health Technol Assess Ser. 2014 Oct 1;14(11):1-32. eCollection 2014. PMID 26330893